CLINICAL TRIAL: NCT06788821
Title: Prenatal Ultrasonographic Assessment of Fetal Thyroid in Patients With Thyroid Pathology
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: FETAL THYROID
Record Dates: First submitted 2024-12-03; First posted 2025-01-23 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-10

CONDITIONS: Thyroid Disease Pregnancy
Keywords: fetal thyroid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Low obstetric risk: i.e., pregnancy with a regular course and not complicated by maternal and/or fetal pathology
  Interventions: Diagnostic Test: Description of the trend of major thyroid ultrasound biometric parameters
- Hypertyroidism: Group con participants with hypertyroidism
  Interventions: Diagnostic Test: Description of the trend of major thyroid ultrasound biometric parameters
- Hypothyroidism: Group of participants with hypothyroidism
  Interventions: Diagnostic Test: Description of the trend of major thyroid ultrasound biometric parameters

INTERVENTIONS:
Diagnostic Test: Description of the trend of major thyroid ultrasound biometric parameters — Use of prenatal ultrasonography for diagnosis and prognostic guidance in suspected fetal thyroid changes.

SUMMARY:
The goal of this observational study is to evaluate the possibility to use prenatal ultrasonography for diagnosis and prognostic guidance in cases of suspected fetal thyroid changes in fetuses belonging to women with thyroid disease and women with low obstetric risk (i.e., pregnancy not complicated by maternal and/or fetal pathology) between 14 and 37 gestational weeks.

The main question it aims to answer is:

Is it possible to diagnose thyroid disease in fetuses early using measurable parameters of the fetal thyroid through ultrasonography?

DETAILED DESCRIPTION:
Current knowledge about fetal thyroid anatomy and the association between ultrasonographic alterations and maternal thyroid disease is not yet comprehensive. A number of observational studies have been conducted describing the possible changes found in fetal thyroid parenchyma in mothers with dysthyroidism. In addition, there are interventional studies that have attempted to modulate anti-thyroid therapy in hyperthyroid mothers depending on the ultrasound changes of the fetal thyroid found. However, to date, the possibility of ultrasound study of the fetal thyroid has not been established, and there are no universally recognized reliable nomograms for the assessment of fetal thyroid biometry.

The present study will provide more information about the possibility to use prenatal ultrasonography for diagnosis and prognostic guidance in cases of suspected fetal thyroid changes. In the latter case, we will be able to more accurately delineate the indication for serious prenatal ultrasound checks, guide counseling with the parental couple, addressing them to possible consultation with pediatric specialist.

Women will be asked to undergo a single ultrasound scan, as per normal clinical practice. With the ultrasound scan it will also be possible to assess parameters that will allow the study of the biometry, morphology and volume of fetal thyroid.

ELIGIBILITY:
Inclusion Criteria:

* Participants between 14 and 37 gestational weeks, who will be followed for the entire period of pregnancy, up to delivery, at the same enrolling center
* Obtaining informed consent for participation in the study
* Maternal age between 18 and 45 years (extremes included)
* Participants with good understanding of the Italian language

Exclusion Criteria:

* Smoking participants
* Patients with BMI>30
* Absence of correct dating of pregnancy within the first trimester
* Pathological conditions (e.g., malabsorptive or socioeconomic conditions that may interfere with fetal growth)
* Twin pregnancy
* Only for the low obstetric risk group of patients: Fetus with malformative pathology

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients from 14 to 37 weeks of pregnancy, with thyroid disease or at low obstetric risk who will undergo obstetric ultrasound at the outpatient clinics of the hospitals where they will deliver.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Fetal thyroid volume = (π/6) × Longitudinal diameter × Antero-Posterior diameter × Transverse diameter (mm3) | Between 14 and 37 pregnancy weeks
  Description of the trend of major thyroid ultrasound biometric parameters in fetuses belonging to women with thyroid disease and women at low obstetrical risk
Right and left thyroid lobe transverse diameter (mm) | Between 14 and 37 pregnancy weeks
  Description of the trend of major thyroid ultrasound biometric parameters in fetuses belonging to women with thyroid disease and women at low obstetrical risk
Longitudinal diameter right and left thyroid lobe (mm) | Between 14 and 37 pregnancy weeks
  Description of the trend of major thyroid ultrasound biometric parameters in fetuses belonging to women with thyroid disease and women at low obstetrical risk
Antero-posterior diameter right and left thyroid lobe (mm) | Between 14 and 37 pregnancy weeks
  Description of the trend of major thyroid ultrasound biometric parameters in fetuses belonging to women with thyroid disease and women at low obstetrical risk

CONTACTS AND LOCATIONS:
Overall Officials: Elena Contro, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (2):
- Italy (2):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna
  - Ospedale Santa Chiara - Trento, Trento, Italy